CLINICAL TRIAL: NCT05375695
Title: Feasibility of Time-Restricted Eating in the Treatment of Type 2 Diabetes - the RESET2 Pilot Study
Brief Title: Feasibility of Time-Restricted Eating in the Treatment of Type 2 Diabetes
Acronym: RESET2pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristine Færch (Other)
Collaborators: Hvidovre University Hospital (Other); University of Leeds (Other); Salk Institute for Biological Studies (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Kristine Færch, Professor and Research Leader, PhD, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-21041830
Record Dates: First submitted 2022-03-27; First posted 2022-05-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes
Keywords: time-restricted eating; type 2 diabetes; obesity; overweight; fasting; circadian rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting; Obesity; Overweight; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-restricted eating (Experimental): Time-restricted eating for 12 weeks (n=20).
  Interventions: Other: Time-restricted eating

INTERVENTIONS:
Other: Time-restricted eating — The intervention consists of an 8-week strict time-restricted eating period, where participants follow the same 10-hour eating window (self-selected timing from 6 am to 8 pm) each day with minimal support to obtain lived experiences with challenges associated with time-restricted eating. Followed by an individually adjusted 4-week time-restricted eating period, including supporting components.
  Staff will help participants select a time-interval that fits into their daily life. Diet is ad libitum and with no further dietary restrictions. The time-restricted eating intervention is an addition to standard care.

SUMMARY:
The overall aim of this pilot study is to examine feasibility of a 12-week 10-hour time-restricted eating intervention in individuals with overweight or obesity and type 2 diabetes. The results of the pilot study will inform recruitment, design and delivery of a future long-term time-restricted randomized controlled trial.

DETAILED DESCRIPTION:
In people with type 2 diabetes (T2D), weight loss is associated with improved glycaemic control and markers of cardiometabolic function as well as reduced use of antidiabetic medicine. Beyond pharmacological treatments, current strategies to reduce body weight and improve glycaemia include energy-restricted diets and increased physical activity.

Lifestyle interventions are complex, affecting many aspects of peoples' daily life. Dietary restrictions often result in rapid weight loss, but the weight is gradually regained by many. Barriers to implement and maintain dietary changes include lack of knowledge, support, and insights into the type and amount of foods eaten. Previous lifestyle interventions targeting weight loss in T2D show efficacy for improving markers of metabolic risk, including weight and glycaemia during the intervention, but relapse of behavior and weight regain are often present.

One reason may be that the intervention is not modified according to the needs of the target group. Often, weight loss interventions are shaped by a 'one size fits all' model where both individual capabilities and motivation as well as social and contextual factors are more or less ignored. A user-based design will facilitate enrolment of participants and likely promote uptake and maintenance of the intervention among participants.

Intermittent fasting regimens have been suggested as efficient strategies for improving cardiometabolic health to a greater extent than can be attributed to the reduction in energy intake alone. Time-restricted eating limits the time available for food intake to typically 4-10 hours/day without other dietary restrictions and has been put forward as a novel, acceptable, and safe lifestyle modification and has shown promising effects on body weight, glucose metabolism, appetite, and cardiometabolic health in individuals at high risk of T2D.

The overall aim of this pilot study is to examine feasibility of a 12-week 10-hour time-restricted eating based intervention in individuals with overweight or obesity and T2D. Participants will attend visit 1 (baseline), visit 2 (8 weeks after baseline) and visit 3 (12 weeks after baseline). The study consists of 8 weeks of strict time-restricted eating, followed by 4 weeks of individually adjusted time-restricted eating.

Specific aims are:

1. To assess adherence and participants' experiences, needs and barriers with an 8-week strict time-restricted eating period, followed by a 4-week period with an individually adjusted time-restricted eating based intervention
2. To examine whether intervention components are delivered by health care professionals as intended
3. To explore if intervention support components are acceptable, useful and sufficient for the participants
4. To study recruitment processes and retention, and related barriers and facilitators
5. To evaluate examination days

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years
* Overweight or obesity (BMI ≥25 kg/m2)
* T2D with HbA1c >53 mmol/mol
* Habitual eating window ≥12 h/day (incl. foods/snacks and energy-containing beverages)
* Associated with the T2D clinic at Steno Diabetes Center Copenhagen (SDCC) or Hvidovre Hospital

Exclusion Criteria:

* Weight loss >5kg last 3 months
* Bariatric surgery or planned bariatric surgery within study duration
* Use of fast acting insulin and combination insulin products
* Unable or unwilling to adhere to time-restricted eating; for instance, due to competing medical conditions.
* A wish to adhere to Ramadan
* For women: current/planned pregnancy or lactation
* Alcohol or drug abuse (judged by investigator) or treatment with disulfiram
* Severe hypoglycaemia within last year (Severe hypoglycaemia, as defined by the American Diabetes Association, denotes severe cognitive impairment requiring external assistance for recovery)
* Inability to understand written and oral information in Danish.
* Diagnosed with an eating disorder in the past 3 years
* Medical condition which, based on investigators assessment, challenges participation including but not limited to severe heart, vascular or lung disease, cancer, chemotherapy, psychiatric gastrointestinal, rheumatic or endocrine diseases etc.
* Concomitant participation in other intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Adherence (%) | Registered 1 day/week on random days per e-mail from baseline to week 8.
  Self-reported adherence to a 10-hour eating window/day during a 8-week strict time-restricted eating period. % compliance = (number of days compliant/total days) * 100%.
Adherence (%) | Registered 1 day/week on random days per e-mail from week 8 to week 12.
  Self-reported adherence to a 10-hour eating window during a 4-week individually adjusted time-restricted eating period. % compliance = (number of days compliant/total days) * 100%.
Participants' experiences, needs and barriers | 8 weeks after baseline.
  Analysis of conversations at visit 2 to assess participants' experiences, needs and barriers with a 8-week strict time-restricted eating period.
Participants' experiences, needs and barriers | 12 weeks after baseline.
  Analysis of interviews at visit 3 to assess participants' experiences, needs and barriers with a 4-week individually adjusted time-restricted eating period, including to explore if intervention support components are acceptable, useful and sufficient for the participants.

SECONDARY OUTCOMES:
Recruitment process and retention | Up to 12 weeks.
  Registered numbers of: people with interest in the project, people attending pre-screening and screening, included participants, drop-outs and completers.
Evaluation of examination days | Interviews at baseline and after 8 and 12 weeks.
  Analysis of interviews to evaluate examination days.
Fidelity | Conversations at baseline and after 8 weeks.
  Assessment of the extent (%) to which the conversations are conducted according to the conversation guidelines. Average score for conversations at baseline and average score for conversations at visit 2 will be calculated.
Body weight (kg) | Measured at baseline and after 8 and 12 weeks
  Measured on a digital scale. Fasted state at baseline and after 12 weeks, non-fasted state after 8 weeks
Body mass index (kg/m^2) | Measured at baseline and after 8 and 12 weeks.
  Calculated from body weight (kg) and height (m). Fasted state at baseline and after 12 weeks, non-fasted state after 8 weeks.
Fat mass (kg) | Measured at baseline and after 12 weeks.
  Measured by electronical bioimpedance. Fasted state at both visits.
Fat free mass (kg) | Measured at baseline and after 12 weeks.
  Measured by electronical bioimpedance. Fasted state at both visits.
Fat percentage (%) | Measured at baseline and after 12 weeks.
  Measured by electronical bioimpedance. Fasted state at both visits.
Waist circumference (cm) | Measured at baseline and after 12 weeks.
  Measured using tape measure.
Hip circumference (cm) | Measured at baseline and after 12 weeks.
  Measured using tape measure.
HbA1c (mmol/mol and %) | Measured at baseline and after 12 weeks.
  Assessed from blood samples in fasted state.
Systolic blood pressure (mmHg) | Measured at baseline and after 12 weeks.
  Measured under resting and fasting conditions.
Diastolic blood pressure (mmHg) | Measured at baseline and after 12 weeks.
  Measured under resting and fasting conditions.
Heart rate (bpm) | Measured at baseline and after 12 weeks.
  Measured under resting and fasting conditions during measurements of blood pressure.
Metabolites | Measured at baseline and after 12 weeks.
  Fasting concentrations of glucose, cholesterols, triglycerides.
Hormone | Measured at baseline and after 12 weeks.
  Fasting concentration of insulin.
Marker of kidney function - Sodium | Measured at baseline and after 12 weeks.
  Fasting concentration of sodium.
Marker of kidney function - Potassium | Measured at baseline and after 12 weeks.
  Fasting concentration of potassium.
Marker of kidney function - Creatinine | Measured at baseline and after 12 weeks.
  Fasting concentration of creatinine.
Markers of kidney function - eGFR | Measured at baseline and after 12 weeks.
  Estimated glomerular filtration rate (eGFR).
Subjective appetite | Measured at baseline and after 12 weeks.
  Rated using visual analogue scales and includes sensations of: Hunger, fullness, satiety, prospective food consumption, wellbeing, nausea, thirst, desire to eat meat, salty, and sweet. The scale range is 0-100 and each end represent the extremes e.g. hunger rating: "I am not hungry at all" to "I have never been this hungry before".
Food choice | Measured at baseline and after 12 weeks.
  Food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Food choice is determined based on frequency of selection made within each food category. The scores range from 0-48 i.e. 0 = foods within a specific food category have not been selected at all to 48 = foods within a specific food category have been selected 48 times.
Implicit wanting | Measured at baseline and after 12 weeks.
  Implicit wanting of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Implicit wanting is assessed based on food choice and response time for selected and non-selected food items as well as mean response time.
Explicit liking | Measured at baseline and after 12 weeks.
  Explicit liking of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Explicit liking is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how pleasant would it be to taste this food right now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Explicit wanting | Measured at baseline and after 12 weeks.
  Explicit wanting of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Explicit wanting is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how much do you want some of this food now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Self-reported physical activity | Measured at baseline and after 12 weeks.
  Assessed from questionnaire International Physical Activity Questionnaire, and measures health-related physical activity. To calculate MET minutes a week multiply the MET value given by the minutes the activity was carried out and again by the number of days that that activity was undertaken.
Self-reported sleep quality | Measured at baseline and after 12 weeks
  Assessed from the questionnaire Pittsburgh Sleep Quality Index. The questionnaire consists of 19 items. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Self-reported health and wellbeing | Measured at baseline and after 12 weeks.
  Assessed from the questionnaire Self-reported Health (SF-12 health survey). SF-12 consists of 12 items. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. A score of 50 or less on the Physical Component Summary has been recommended as a cut-off to determine a physical condition; while a score of 42 or less on the Mental Component Summary may be indicative of 'clinical depression'.
Self-reported sleepiness | Measured at baseline and after 12 weeks.
  Assessed from the questionnaire the Epworth Sleepiness Scale. The questionnaire consists of 8 questions, which is weighted on a 0-3 interval scale. A low total score can be interpreted as a normal daytime sleepiness, and a higher score as a mild, moderate and severe excessive daytime sleepiness, respectively.
Self-reported chronotype | Measured at baseline and after 12 weeks.
  Assessed from the questionnaire Munich Chronotype Questionnaire (MCTQ). The questionnaire consists of 17 questions to identify type of chronotype. The MCTQ uses the midpoint between sleep on- and offset on free days (mid-sleep on free days) to assess chronotype.
Self-reported food intake | Measured at baseline and after 12 weeks
  Assessed from questionnaire Food Frequency Questionnaire. The questionnaire collects dietary data and uses a context-specific food list to estimate the usual diet. The questionnaire consists of 15 items with sub questions. Output is total energy intake and macronutrient composition.
Self-reported night eating | Measured at baseline and after 12 weeks.
  Assessed from questionnaire The Night Eating Questionnaire. The questionnaire consists of 14 items, that can be rated from 0 to 4. All items except item 13 are summed to obtain a global score. A total score ≥ 25 has been proposed as a lenient threshold for night eating syndrome.
Self-reported eating behavior | Measured at baseline and after 12 weeks.
  Assessed from questionnaire The Dutch Eating Behavior Questionnaire. It consists of 33 items and comprises three scales that measure emotional, external and restrained eating.Items can be rated from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
Self-reported control over eating | Measured at baseline and after 12 weeks.
  Assessed from the questionnaire Control over Eating Questionnaire. It comprises 21 items designed to assess the intensity and type of food cravings an individual experiences, as well as subjective sensations of appetite and mood. Each item can be rated from 1 to 5 on a continuous scale. a lower scale. A higher score indicate less control over eating.
Self-reported fatigue/tiredness | Measured at baseline and after 12 weeks.
  Assessed from questionnaire Fatigue Assessment Scale (FAS). The questionnaire consists of 10 items. Each item can be rated from 1 to 5. The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
Self-reported information on social relations and support | Measured at baseline and after 12 weeks.
  Assessed from 8 selected items on social relations and support from The Danish National Health Survey. Item 1-7 provides information on how often a person is in contact with other people (family, husband/wife, partners, friends, neighbors, etc.), and can be rated from 'daily or almost daily', 'once or twice weekly', 'once or twice monthly', 'less than once monthly' to 'never'. Item 8 provides information on whether a person has somebody to talk to if he/she has problems or needs support, and can be rated 'yes, always', 'yes, mostly', 'yes, sometimes', and 'no, never or almost never'.
Self-reported diabetes distress | Measured at baseline and after 12 weeks.
  Assessed from the Problem Areas in Diabetes Scale (PAID-5 scale) comprising five of the emotional-distress questions of the full PAID items. Each item can be rated from 0 to 4. A total score of ≥ 8 indicates possible diabetes related emotional distress.
Self-reported well-being | Measured at baseline and after 12 weeks
  Assessed from the WHO (Five) Well-being Index. The WHO-5 consists of five statements, which respondents rate from 0 to five (in relation to the past two weeks).The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Self-reported diabetes management | Measured at baseline and after 12 weeks.
  Assessed from 9 selected items on diabetes management from the The Danish National Patient Reported Outcome Questionnaire, version 1.05. The items can be rated from 'very sure/confident' to 'not sure/confident at all'.
Sexual satisfaction | Measured at baseline and after 12 weeks.
  Assessed from 1 item on sexual satisfaction from the questionnaire The Danish National Health Survey. The item addresses to which degree a persons sexual needs are covered. The item can be rated from 'to a very high degree' to 'not at all'.
Sexual functioning | Measured at baseline and after 12 weeks.
  Assessed from 4 items on sexual functioning from the Danish National Patient Reported Outcome Questionnaire, version 1.05. Item 1 can be rated 'yes' or 'no'. 'Yes' represents problems with sexual functioning. Item 2-4 can be rated from 'not at all' to 'extreme', where extreme represents problems with sexual functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Færch, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Termannsen AD, Bjerre N, Hansen GS, Jalking L, Faerch K, Hempler NF, Quist JS, Varming A. Theory-based process evaluation of a non-randomised single-arm pilot study investigating time-restricted eating in the treatment of type 2 diabetes-the RESET2 pilot study. Pilot Feasibility Stud. 2025 Nov 6;11(1):135. doi: 10.1186/s40814-025-01715-4. PMID 41199408